CLINICAL TRIAL: NCT06841003
Title: Laparoscopic Antibiotic Lavage to Prevent Intra-abdominal Abscess Formation in Complicated Appendicitis (ALPACA), a Multicenter Single-blinded RCT.
Brief Title: Laparoscopic Antibiotic Lavage to Prevent Intra-abdominal Abscess Formation in Complicated Appendicitis
Acronym: ALPACA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Spaarne Gasthuis (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-514850-59-00
Record Dates: First submitted 2025-02-03; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Complicated Appendicitis; Intra-Abdominal Abscess
MeSH Terms: conditions — Abdominal Abscess | interventions — Gentamicins; Clindamycin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laparoscopic antibiotic lavage (Experimental)
  Interventions: Drug: Laparoscopic antibiotic peritoneal lavage with gentamicin / clindamycin
- Control group (No Intervention)

INTERVENTIONS:
Drug: Laparoscopic antibiotic peritoneal lavage with gentamicin / clindamycin — Peritoneal antibiotic lavage using a solution of gentamicin/clindamycin in NaCl 0.9%.
  Arms: Laparoscopic antibiotic lavage

SUMMARY:
Appendicitis is one of the most common causes of acute surgical admission. Presently, two types of appendicitis are distinguished: complicated and uncomplicated (phlegmonous). Complicated appendicitis (CA) is defined as gangrenous and/or perforated appendicitis and/or appendicitis with an intra-abdominal or pelvic abscess. Laparoscopic appendectomy has become the preferential mode of surgical treatment. However, development of an intra-abdominal abscess (IAA) remains an important and clinically relevant complication following appendectomy, especially in complicated appendicitis. Although patients with complicated appendicitis receive postoperative intravenous antibiotics, the incidence of IAA remains considerable. The reported incidence of IAA in children and adults with CA is 7.9% - 24%. We recently reported an IAA rate of 12.3% after laparoscopic appendectomy for CA in our own institution. Patients with IAA are readmitted and treated with either antibiotics, image-guided percutaneous drainage, surgical reintervention, or a combination of these treatments. Furthermore, IAA represents a considerable burden for the healthcare system with high readmission rates and reinterventions, prolonged hospital stay, and therefore increased medical costs. Intra operative techniques aiming at more effective infection source control represent a clinically relevant area of investigation. Laparoscopic antibiotic lavage represents a promising concept in order to reduce intra-abdominal abscess formation. Antibiotic lavage is mainly known for the treatment of peritoneal dialysis associated peritonitis. Several studies show promising results of antibiotic peritoneal lavage on the incidence of surgical site infections (SSIs) including IAA in patients with CA. However, these studies were retrospective or conducted in a small number of patients who underwent an open appendectomy while high quality randomized controlled trials have not been performed yet.

The aim of the ALPACA study is to evaluate the effect of laparoscopic antibiotic peritoneal lavage with gentamicin / clindamycin for 3 minutes after appendectomy on the incidence of IAA in patients with CA.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 8 years with a preoperative diagnosis of acute appendicitis either with or without clinical or radiological suspicion of CA undergoing a laparoscopic appendectomy for intra-operative confirmed CA that can provide a signed written consent form.

Exclusion Criteria:

* Age under 8 years;
* Not able to give informed consent (language barrier, legally incapable)
* Any contraindication for the use of the study medication:

  * Hypersensitivity to clindamycin or to any of the excipients benzyl alcohol, sodium edetate, water, or to lincomycin;
  * Hypersensitivity to gentamicin or to sodium metabisulfite: particularly in asthmatic patients, this may trigger bronchospasms and anaphylactic shock or to any of the excipients: disodium edetate, sodium hydroxide, sodium metabisulfite (E223), water for injections;
* Severe sepsis defined as sepsis-induced tissue hypoperfusion or organ dysfunction that includes any of the following thought to be caused by the infection:

  * Sepsis-induced hypotension
  * Lactate above upper limits laboratory normal
  * Urine output <0.5 mL/kg/h for more than 2h despite adequate fluid resuscitation
  * Acute lung injury with PaO2/FiO2 <250 in the absence of pneumonia as infection source
  * Acute lung injury with PaO2/FiO2 <200 in the presence of pneumonia as infection source
  * Creatinine >2.0 mg/dL (176.8 μmol/L)
  * Bilirubin >2mg/dL (34.2 μmol/L)
  * Platelet count < 100,000 μL
  * Coagulopathy (international normalized ratio (INR) > 1.5);
* ASA IV score;
* Known malignancy;
* Renal dysfunction (i.e. eGFR ≤ 60);
* Immunocompromised patients (i.e. hematological malignancies, HIV/AIDS, bone marrow transplantation, splenectomy, genetic disorders such as severe combined immunodeficiency, chemotherapy, dialysis, solid organ transplant, and immunosuppressant use (such as corticosteroids in patients with rheumatoid arthritis));
* Pregnancy;
* Known allergies to either gentamicin or clindamycin;
* Known colonization of bacteria resistant to either gentamicin or clindamycin;

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 752 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The incidence of intra-abdominal abscess (IAA) | Within 30 days follow-up

SECONDARY OUTCOMES:
The number of participants with wound infections measured by tracking any wound complications that these patients have and comparing the incidence between treatment arms | Within 90-days follow-up
The type of treatment for the intra-abdominal abscess, consisting of percutaneous (radiological drainage), surgical drainage, antibiotic treatment or observation only | Within 90-days follow-up
Microbial cultures of intra-operative aspirate, based on cultures | Within 90-days follow-up
Operating time | From the moment of start surgery (the incision) to wound closure.
Readmission rate | Within 90-days follow-up
Reoperation rate | Within 90-days follow-up
Length of stay (including readmission) | Within 90-days follow-up
Adverse events of antibiotic peritoneal lavage | Within 90-days follow-up
Surgical complications according to the Clavien-Dindo classification | Within 90-days follow-up
Mortality | Within 90-days follow-up
Quality of life | Within 90-days follow-up
  Measured by digital questionnaire of EuroQol-5 Dimension (EQ-5D)
The number of postoperative consultations will be measured by tracking any postoperative consultation that these patients have and comparing the incidence between treatment arms | Within 90-days follow-up
  Including emergency department visits, telephone consultations and outpatient consultations
Cost-effectivity, | Within 90-days follow-up
  Cost-effectivity will be determined by IMTA Productivity Cost Questionnaire (iPCQ)
Microbial cultures of postoperative intra-abdominal asbcess, based on cultures | Within 90-days follow-up
Cost-effectivity | Within 90-days follow-up
  The cost-effectivity will be determined by iMTA Medical Consumption Questionnaire